CLINICAL TRIAL: NCT01955070
Title: Use of a Multimedia Presentation to Enhance the Informed Consent for Ketamine Sedation in a Pediatric Emergency Department
Brief Title: Use of a Multimedia Presentation for Informed Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Sandra Spencer, Assistant Professor of Clinical Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MMP for Informed Consent
Record Dates: First submitted 2013-09-03; First posted 2013-10-07 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Improving Informed Consent Process
Keywords: Informed consent; Ethics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Implementation (Experimental): Multimedia Presentation for Ketamine sedation
  Interventions: Other: Multimedia Presentation for Ketamine sedation
- Intervention (Experimental): Multimedia Presentation for Ketamine sedation
  Interventions: Other: Multimedia Presentation for Ketamine sedation
- Control (No Intervention): Patients that received the standard consent with signed consent form

INTERVENTIONS:
Other: Multimedia Presentation for Ketamine sedation — PowerPoint presentation created with approval of section of emergency medicine for informed consent for ketamine sedation
  Arms: Implementation; Intervention

SUMMARY:
This is a prospective cohort study in which the standard verbal informed consent process for ketamine sedation is compared to a multimedia informed consent process. The goals include determining if parents prefer a multimedia consent process and evaluating the effectiveness of multimedia consent process.

DETAILED DESCRIPTION:
BACKGROUND: Informed consent (IC) is an ethical process for ensuring patient autonomy. Multimedia presentations (MMP) often aid the IC process for research studies. Thus, it follows that MMP would improve IC in clinical settings.

OBJECTIVE: To determine if MMP for the IC process for ketamine sedation improves parental satisfaction and comprehension as compared to standard practice.

DESIGN/METHODS: This two phase study compared two methods of IC for ketamine sedation of pediatric patients. Phase one was a randomized, prospective study that compared the standard verbal consent to a MMP. Phase two implemented the MMP into daily work flow. Parents completed a survey evaluating their satisfaction of the IC process and assessing their knowledge of ketamine sedation. Primary outcome measures were parental overall satisfaction with the IC process and knowledge of ketamine sedation.

ELIGIBILITY:
Inclusion Criteria:

* Receiving ketamine sedation for fracture reduction
* Less than 18 years of age
* English as primary language

Exclusion Criteria:

* patients who received medications in addition to ketamine for sedation
* Families where English was not the primary language

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Parents' satisfaction with the informed consent process | Within 1 hour of consent
  Parents are given a survey with a 5-point Likert scale to evaluated their satisfaction with the informed consent process
The parent's knowledge of ketamine sedation. | Within one hour of consent
  The parents are give a multiple choice quiz on the information present on ketamine sedation

SECONDARY OUTCOMES:
Satisfaction within each domain | Within one hour of consent
  The satisfaction questions on the survey are divided into groups addressing the four key elements of informed consent: beneficence, maleficence, content, and assent.
Comparison of satisfaction and knowledge with demographics | Within one hour of consent
  The survey and quiz results are compared depending on demographics
Provider Satisfaction | Time 0 and 6 months later
  Provider satisfaction was collected using a Likert scale at the time the presentation was embedded into the computer order entry system. They were re-surveyed 6 months later to see if there was any change in the satisfaction results

CONTACTS AND LOCATIONS:
Overall Officials: Sandra P Spencer, MD, Principal Investigator — Nationwide Childrens, Department of Emergency Medicine
Locations (1):
- Nationwide Childrens, Columbus, Ohio, United States

REFERENCES:
- [Background] Akkad A, Jackson C, Kenyon S, Dixon-Woods M, Taub N, Habiba M. Informed consent for elective and emergency surgery: questionnaire study. BJOG. 2004 Oct;111(10):1133-8. doi: 10.1111/j.1471-0528.2004.00240.x. PMID 15383117
- [Background] Baren J, Campbell CF, Schears RM, Shofer FS, Datner EM, Hollander JE. Observed behaviors of subjects during informed consent for an emergency department study. Ann Emerg Med. 2010 Jan;55(1):9-14. doi: 10.1016/j.annemergmed.2009.09.023. Epub 2009 Nov 22. PMID 19931940
- [Background] Agre P, Rapkin B. Improving informed consent: a comparison of four consent tools. IRB. 2003 Nov-Dec;25(6):1-7. No abstract available. PMID 15035248
- [Background] Flory J, Emanuel E. Interventions to improve research participants' understanding in informed consent for research: a systematic review. JAMA. 2004 Oct 6;292(13):1593-601. doi: 10.1001/jama.292.13.1593. PMID 15467062
- [Background] Nwomeh BC, Hayes J, Caniano DA, Upperman JS, Kelleher KJ. A parental educational intervention to facilitate informed consent for emergency operations in children. J Surg Res. 2009 Apr;152(2):258-63. doi: 10.1016/j.jss.2008.01.008. Epub 2008 Feb 4. PMID 18374948
- [Derived] Spencer SP, Stoner MJ, Kelleher K, Cohen DM. Using a Multimedia Presentation to Enhance Informed Consent in a Pediatric Emergency Department. Pediatr Emerg Care. 2015 Aug;31(8):572-6. doi: 10.1097/PEC.0000000000000513. PMID 26221786